CLINICAL TRIAL: NCT04717947
Title: Interval Between Neoadjuvant Therapy and Surgery in the Treatment of Locally Advanced Rectal Cancer
Brief Title: Interval Between Neoadjuvant Therapy and Surgery in the Treatment of Locally Advanced Rectal Cancer (CRONOS)
Acronym: CRONOS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Complejo Hospitalario Universitario de Santiago (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital de Sant Joan Despí Moisès Broggi (Other); Hospital del Mar (Other); Hospital Son Espases (Other); Hospital Universitario La Fe (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Fundacion del Hospital Nacional de Paraplejicos para la Investigacion y la Integracion (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2019/1109
Record Dates: First submitted 2020-10-02; First posted 2021-01-22 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-10

CONDITIONS: Rectal Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Short interval group: ≤ 8weeks between the end of neoadjuvant therapy and surgery
  Interventions: Procedure: Interval between NAT and surgery
- Intermediate interval group: > 8 and ≤ 12 weeks between the end of neoadjuvant therapy and surgery
  Interventions: Procedure: Interval between NAT and surgery
- Long interval group: > 12 weeks between the end of neoadjuvant therapy and surgery

INTERVENTIONS:
Procedure: Interval between NAT and surgery — Evaluate three groups according to the interval between the end of neoadjuvant therapy and surgery.
  Groups: Intermediate interval group; Short interval group

SUMMARY:
The investigators evaluate the response of rectal cancer to neoadjuvant therapy and classify the response according to specific periods of time after the end of neoadjuvant treatment.

DETAILED DESCRIPTION:
In the treatment of locally advanced rectal cancer, an optimal interval between neoadjuvant therapy and surgery might improve oncological outcomes. Besides, those patients who achieve a good response might benefit from active surveillance, avoiding surgical comorbidities. This optimal interval is yet to be defined. This study will aim to better define the role of time interval between the end of neoadjuvant therapy (NAT) and TME in Spanish regions, together with analyzing the importance of restaging MRI and define the basis for implementing a "watch and wait" protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients suitable for elective surgical resection of biopsy-confirmed rectal adenocarcinoma (0-15 cm from the anal verge) determined by rectal cancer protocol magnetic resonance imaging.
* Patients treated with long-course neoadjuvant chemoradiotherapy (nCRT).
* Patients treated with short-course radiotherapy with delayed surgery.
* Clinical stage IIA, IIB, IIIA, IIIB, IIIC (cT3/cT4, or cN1/cN2 with any cT, M0) determined by rectal cancer protocol magnetic resonance imaging

Exclusion Criteria:

* Intolerance or contraindication to planned NAT.
* Patients who have not finished NAT for any reason.
* Patients with unknown cT or cM.
* Tumors previously treated with local excision or with distant metastatic disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a national multicentre retrospective cohort study. Participating centres are tertiary referral hospitals from different Spanish regions, which agreed to enter information in a standardized database, of all patients in their institute who had biopsy-confirmed rectal adenocarcinoma and had received neoadjuvant therapy. All patients with low, mid and high rectal cancer (0-15 cm from the anal verge), at a clinical stage IIA, IIB, IIIA, IIIB, IIIC (cT3/cT4, or cN1/cN2 with any cT, M0) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2021-06-25 (Estimated)

PRIMARY OUTCOMES:
Pathological response | 2000-2019
  Grade as complete
Circumferential margin (CRM) | 2000-2019
  Described as free (CRM >1 mm)
Distal resection margin (DRM) | 2000-2019
  Described as free (DRM >1 mm)
Quality of the specimen | 2000-2019
  Described as complete or incomplete

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lacy, PhD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No